CLINICAL TRIAL: NCT02256631
Title: Open-Label, Dose-Escalating, Phase I Study to Determine Safety and Pharmacokinetic Parameters of Subcutaneous (SC) VRC01, VRC01LS, and VRC07-523LS, Potent Anti-HIV Neutralizing Monoclonal Antibodies, in HIV-1-Exposed Infants
Brief Title: Evaluating the Safety and Pharmacokinetics of VRC01, VRC01LS, and VRC07-523LS, Potent Anti-HIV Neutralizing Monoclonal Antibodies, in HIV-1-Exposed Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMPAACT P1112; 11903 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Dose Group 1 (Experimental): Infants in Dose Group 1 received a single VRC01 20 mg/kg injection less than 72 hours after birth.
  Interventions: Biological: VRC01
- Dose Group 2 (Experimental): Infants in Dose Group 2 received a single VRC01 40 mg/kg injection less than 72 hours after birth.
  Interventions: Biological: VRC01
- Dose Group 3 (Experimental): Infants in Dose Group 3 received a VRC01 40 mg/kg injection less than 5 days after birth. They then received a VRC01 20 mg/kg injection monthly for at least 6 months and no more than 18 months while breastfeeding.
  Interventions: Biological: VRC01
- Dose Group 4, Cohort 1 (Experimental): Infants in Cohort 1 received a single VRC01LS injection less than 72 hours after birth. Dose was based on weight: 80 mg for infants weighing less than 4.5 kg and 100 mg for infants weighing 4.5 kg or greater.
  Interventions: Biological: VRC01LS
- Dose Group 4, Cohort 2 (Experimental): Infants in Cohort 2 received an initial VRC01LS injection no longer than 5 days after birth. Dose was based on weight: 80 mg for infants weighing less than 4.5 kg and 100 mg for infants weighing 4.5 kg or greater. A second dose of 100 mg VRC01LS was administered at Week 12 if an infant was still breastfeeding.
  Interventions: Biological: VRC01LS
- Dose Group 5, Cohort 1 (Experimental): Infants in Cohort 1 received a single VRC07-523LS injection less than 72 hours after birth. Dose was based on weight: 80 mg for infants weighing less than 4.5 kg and 100 mg for infants weighing 4.5 kg or greater.
  Interventions: Biological: VRC07-523LS
- Dose Group 5, Cohort 2 (Experimental): Infants in Cohort 2 received an initial VRC07-523LS injection no longer than 5 days after birth. Dose was based on weight: 80 mg for infants weighing less than 4.5 kg and 100 mg for infants weighing 4.5 kg or greater. A second dose of 100 mg VRC07-523LS was administered at Week 12 if an infant was still breastfeeding.
  Interventions: Biological: VRC07-523LS

INTERVENTIONS:
Biological: VRC01 — Administered by subcutaneous injection in the thigh
  Other Names: VRC-HIVMAB-060-00-AB; VRC01 mAb
  Arms: Dose Group 1; Dose Group 2; Dose Group 3
Biological: VRC01LS — Administered by subcutaneous injection in the thigh
  Other Names: VRC-HIVMAB080-00-AB
  Arms: Dose Group 4, Cohort 1; Dose Group 4, Cohort 2
Biological: VRC07-523LS — Administered by subcutaneous injection in the thigh
  Other Names: VRC-HIVMAB075-00-AB
  Arms: Dose Group 5, Cohort 1; Dose Group 5, Cohort 2

SUMMARY:
The purpose of this study was to assess the safety and pharmacokinetics (PK) of three monoclonal antibodies, VRC01, VRC01LS, and VRC07-523LS, in HIV-exposed infants who are at increased risk of mother-to-child HIV transmission.

DETAILED DESCRIPTION:
VRC01, VRC01LS, and VRC07-523LS are anti-HIV neutralizing monoclonal antibodies that may help prevent mother-to-child transmission of HIV. This study enrolled HIV-infected mothers who were at increased risk of passing HIV on to their children. The purpose of this study was to assess the safety and PK of VRC01, VRC01LS, and VRC07-523LS in HIV-exposed infants.

This study enrolled mother-infant pairs into five dose groups. Infants enrolled in Dose Group 1 and Dose Group 2 received a single VRC01 injection less than 72 hours after birth. Infants in Dose Group 3 received a VRC01 injection less than 5 days after birth, followed by VRC01 injections monthly for at least 6 months and no more than 18 months, while breastfeeding.

Dose Groups 4 and 5 each enrolled infants into two cohorts: Cohort 1 (non-breastfeeding) or Cohort 2 (breastfeeding). Infants in Dose Group 4, Cohort 1 received a single VRC01LS injection less than 72 hours after birth. Infants in Dose Group 4, Cohort 2 received an initial VRC01LS injection no longer than 5 days after birth, and a second VRC01LS injection at Week 12 if they were still breastfeeding. Infants in Dose Group 5, Cohort 1 received a single VRC07-523LS injection less than 72 hours after birth. Infants in Dose Group 5, Cohort 2 received an initial VRC07-523LS injection no longer than 5 days after birth, and a second VRC07-523LS injection at Week 12 if they were still breastfeeding.

The mothers did not receive any VRC01, VRC01LS, or VRC07-523LS injections. At study entry, all mothers underwent a medical history review and a blood collection, and then the study ended for the mothers.

Infants in Dose Groups 1 and 2 attended study visits at days 0, 1, 3, 7, 14, 28 and at weeks 8, 16, 24, and 48. Infants in Dose Group 3 attended study visits at days 0, 1, 14, 28 and at weeks 8, 12, 16, 20, 24, and every 4 weeks until cessation of breastfeeding or week 72, then at weeks 84 and 96. Infants in Dose Group 4 attended study visits at days 0, 1, 14, 28 and at weeks 8, 12, 24, 36, 48, 60, 72, 84 and 96, with additional visits at weeks 14 and 16 for Cohort 2 participants. Infants in Dose Group 5 attended study visits at days 0, 1, 3, 7, 14, 28 and at weeks 8, 12, 24, 36, 48, 60, 72, 84 and 96, with additional visits at weeks 14 and 16 for Cohort 2 participants. Visits included a medical history review, physical examination, blood collection, and oral fluid collection.

ELIGIBILITY:
Maternal Inclusion Criteria:

* HIV infection
* Greater than or equal to 18 years of age
* Able and willing to provide signed informed consent for herself and her infant

Maternal Exclusion Criteria:

* Prior participation in any HIV-1 vaccine trial
* Receipt of any other active or passive HIV immunotherapy or investigational product during this pregnancy. (Note that administration of Food and Drug Administration [FDA]-approved antiretroviral (ARV) drugs when used to treat disease or prevent mother-to-child transmission were not considered investigational.)
* Documented or suspected serious medical illness or immediate life-threatening condition (other than HIV infection) in the mother that may have interfered with the ability to complete study requirements, as judged by the examining clinician

Infant Inclusion Criteria:

* Born to an HIV-1-infected woman who met all maternal inclusion/exclusion criteria listed above
* Gestational age, by best obstetrical, ultrasound, or infant exam, greater than or equal to 36 weeks
* Birth weight greater than or equal to 2.0 kg
* Allowable infant age at the time of enrollment was dependent on the Dose Group and Cohort:

  * Dose Groups 1, 2, 4 and 5 (Cohort 1): Less than 72 hours of age, and anticipated availability to receive VRC immunization at less than 72 hours after birth.
  * Dose Groups 3, 4 and 5 (Cohort 2): Less than or equal to 5 days of age, and anticipated availability to receive VRC immunization no more than 5 days after birth.
* At increased risk of HIV acquisition defined as documentation of one or more of the following risk factors:
* Dose Groups 1, 2, 4 and 5 (Cohort 1), only:

  * Mother received no antiretroviral therapy (ART) during pregnancy or mother began or reinitiated ART (after an interruption of greater than 14 days), during the third trimester of pregnancy; or
  * Mother with any detectable viral replication (HIV RNA above the limit of detection) at last measurement prior to delivery determined within 30 days of delivery; or
  * Prolonged rupture of membranes (greater than 12 hours); or
  * Mother with documented 2-class resistant HIV infection, which may have included historical documentation of lack of response

    * Women who had a documented history of virologic failure while on non-nucleoside reverse transcriptase inhibitors (NNRTIs) but who had no resistance testing at the time of viral failure were considered to have NNRTI-documented resistance.
* Dose Groups 3, 4 and 5 (Cohort 2), only (African sites):

  * Mother intended to breastfeed

Infant Exclusion Criteria:

* Receipt of any other active or passive HIV immunotherapy or investigational product other than the study vaccine (Note: Infant prophylaxis with any licensed ARV drugs clinically prescribed to prevent mother-to-child HIV transmission were not considered investigational.)
* Receipt of or anticipated need for blood products, immunoglobulin, or immunosuppressive therapy. This included infants who required hepatitis B immunoglobulin (HBIG) but did not require exclusion of infants who received hepatitis B vaccine in the newborn period.
* Documented or suspected serious medical illness, serious congenital anomaly, or immediate life-threatening condition in the infant that may have interfered with the ability to complete study requirements, as judged by the examining clinician
* Any requirement for supplemental oxygen beyond 24 hours of life or requiring supplemental oxygen at the time of the VRC01, VRC01LS, or VRC07-523LS dose
* Baseline laboratory results:

  * Hemoglobin less than 12.0 g/dL
  * Platelet count less than 100,000 cells/mm^3
  * Absolute neutrophil count: for infants less than or equal to 24 hours old, less than 4,000 cells/mm^3; for infants greater than 24 hours old, less than 1,250 cells/mm^3
  * Serum glutamic pyruvic transaminase (SGPT) greater than or equal to 1.25 times upper limit of age adjusted normal
* Dose Groups 1, 2, 4 and 5 (Cohort 1), only: Infant was breastfeeding at time of enrollment or mother had indicated an intention to initiate breastfeeding. Note: if a child was breastfed prior to known maternal diagnosis (in the case of a woman diagnosed in the intrapartum period), the child was still eligible as long as breastfeeding was stopped by the time the child was enrolled and there was no plan to resume breast milk feeding.

Ages: 0 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Coleen Cunningham, MD, Study Chair — Duke University
Locations (14):
- United States (10):
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - Emory University School of Medicine NICHD CRS, Atlanta, Georgia
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Bronx-Lebanon Hospital Center NICHD CRS, The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - Texas Children's Hospital CRS, Houston, Texas
- Puerto Rico (2):
  - San Juan City Hosp. PR NICHD CRS, San Juan, PR
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
- Famcru Crs, Tygerberg, Western Cape, South Africa
- Harare Family Care CRS, Harare, Zimbabwe

REFERENCES:
- [Result] Cunningham CK, McFarland EJ, Morrison RL, Capparelli EV, Safrit JT, Mofenson LM, Mathieson B, Valentine ME, Perlowski C, Smith B, Hazra R, Purdue L, Muresan P, Harding PA, Mbengeranwa T, Robinson LG, Wiznia A, Theron G, Lin B, Bailer RT, Mascola JR, Graham BS; IMPAACT P1112 team. Safety, Tolerability, and Pharmacokinetics of the Broadly Neutralizing Human Immunodeficiency Virus (HIV)-1 Monoclonal Antibody VRC01 in HIV-Exposed Newborn Infants. J Infect Dis. 2020 Jul 23;222(4):628-636. doi: 10.1093/infdis/jiz532. PMID 31681963
- [Result] McFarland EJ, Cunningham CK, Muresan P, Capparelli EV, Perlowski C, Morgan P, Smith B, Hazra R, Purdue L, Harding PA, Theron G, Mujuru H, Agwu A, Purswani M, Rathore MH, Flach B, Taylor A, Lin BC, McDermott AB, Mascola JR, Graham BS; International Maternal Pediatric Adolescent AIDS Clinical Trials Network (IMPAACT) P1112 Team. Safety, Tolerability, and Pharmacokinetics of a Long-Acting Broadly Neutralizing Human Immunodeficiency Virus Type 1 (HIV-1) Monoclonal Antibody VRC01LS in HIV-1-Exposed Newborn Infants. J Infect Dis. 2021 Dec 1;224(11):1916-1924. doi: 10.1093/infdis/jiab229. PMID 34009371
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017) — http://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 mother-infant pairs were enrolled in the study. Since the mothers did not receive any treatment on study and were taken off study immediately after enrollment, the number of participants shown in all tables is the number of infants (83). Participants were enrolled from June 2015 to February 2020, at 14 medical clinics in the United States, Puerto Rico, South Africa and Zimbabwe.
Pre-assignment Details: Dose groups enrolled sequentially. There was no randomization.
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Started | 13 | 14 | 13 | 10 | 11 | 11 | 11
Completed | 12 | 11 | 13 | 6 | 10 | 6 | 7
Not Completed | 1 | 3 | 0 | 4 | 1 | 5 | 4
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Unable to get to clinic | 0 | 2 | 0 | 1 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected only for infants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2 | Total
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11 | 11 | 11 | 83
Age, Customized [Median (Full Range); unit: days]
  Age at first dose | 2 [0 to 3] | 2 [0 to 3] | 2 [1 to 5] | 2 [0 to 3] | 2 [1 to 4] | 1 [1 to 3] | 4 [1 to 5] | 2 [0 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 4 | 6 | 6 | 3 | 37
  Male | 8 | 6 | 8 | 6 | 5 | 5 | 8 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 0 | 1 | 0 | 2 | 0 | 12
  Not Hispanic or Latino | 8 | 10 | 13 | 9 | 11 | 8 | 11 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 11 | 13 | 8 | 11 | 8 | 11 | 68
  White | 6 | 2 | 0 | 2 | 0 | 1 | 0 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  United States | 10 | 9 | 0 | 7 | 0 | 11 | 0 | 37
  South Africa | 1 | 5 | 10 | 3 | 5 | 0 | 7 | 31
  Zimbabwe | 0 | 0 | 3 | 0 | 6 | 0 | 4 | 13
Birth Weight [Median (Full Range); unit: grams] | 3045 [2330 to 4675] | 3160 [2609 to 3580] | 2860 [2330 to 4320] | 2865 [2535 to 4045] | 2920 [2500 to 3545] | 2810 [2528 to 3540] | 3235 [2260 to 4375] | 2920 [2260 to 4675]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died
Description: The Overall Number of Participants Analyzed represents infants. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Deaths from day 0 to 4 weeks after the participants' last immunization were included.
Time Frame: From day 0 to 4 weeks after last immunization (at week 4 for Dose Groups 1, 2, 4-Cohort 1, 5-Cohort 1; at week 16-48 for Dose Group 3; at week 16 for Dose Group 4-Cohort 2, 5-Cohort 2.)
Population: All infant study participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11 | 11 | 11
percentage of participants | 0 [0 to 21] | 0 [0 to 19] | 0 [0 to 21] | 0 [0 to 26] | 0 [0 to 24] | 0 [0 to 24] | 0 [0 to 24]

2. Primary Outcome: Percentage of Participants With an Occurrence of at Least One Grade 3 or Higher Adverse Event (AE)
Description: The Overall Number of Participants Analyzed represents infants. AE severity grading was based on the Division of AIDS (DAIDS) AE Grading table, Corrected Version 2.1. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Adverse events from day 0 to 4 weeks after the participants' last immunization were included.
Time Frame: as for outcome 1
Population: All infant study participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11 | 11 | 11
percentage of participants | 31 [11 to 57] | 14 [3 to 39] | 31 [11 to 57] | 10 [1 to 39] | 27 [8 to 56] | 36 [14 to 65] | 9 [0 to 36]

3. Primary Outcome: Percentage of Participants With at Least One VRC01-, VRC01LS-, or VRC07-523LS-related Grade 3 or Higher Adverse Event (AE)
Description: The Overall Number of Participants Analyzed represents infants. AE severity grading was based on the Division of AIDS (DAIDS) AE Grading table, Corrected Version 2.1. The study sites assessed and determined if AEs were related to study treatment. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Adverse events from day 0 to 4 weeks after the participants' last immunization were included.
Time Frame: as for outcome 1
Population: All infant study participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11 | 11 | 11
percentage of participants | 0 [0 to 21] | 0 [0 to 19] | 0 [0 to 21] | 0 [0 to 26] | 0 [0 to 24] | 0 [0 to 24] | 0 [0 to 24]

4. Primary Outcome: Percentage of Participants Diagnosed With HIV Infection
Description: The Overall Number of Participants Analyzed represents infants. Diagnosis testing was performed using a HIV-1 NAT (nucleic acid testing) by a method that detects DNA. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. HIV diagnoses from day 0 to 4 weeks after the participants' last immunization were included.
Time Frame: as for outcome 1
Population: All infant study participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11 | 11 | 11
percentage of participants | 0 [0 to 21] | 0 [0 to 19] | 0 [0 to 21] | 0 [0 to 26] | 0 [0 to 24] | 0 [0 to 24] | 0 [0 to 24]

5. Primary Outcome: Pharmacokinetics (PK) Parameter: Area Under the Curve (AUC) for Dose Groups 1, 2, 3 and 4
Description: The Overall Number of Participants Analyzed represents infants. PK parameters were determined from plasma concentration-time profiles using noncompartmental methods (SAS 9.4, Cary, NC). AUC0-28 days (area-under-the-curve from 0 to 28 days) for Dose Groups 1, 2 and 3 and AUC0-84 days for Dose Group 4, were determined using the linear trapezoidal rule. Median and range were summarized.
Time Frame: Dose Groups (DG) 1, 2: at days 0, 1, 3, 7, 14, 28; DG 3: at days 0, 1, 14, 28, weeks 16, 20, 24; DG 4-Cohort 1: at days 0, 1, 14, 28; Cohort 2: at days 0, 1, 14, 28, 84.
Population: Infants who received the correct dose and were evaluated for PK at the designated timepoints.
Measure: Median (Full Range); unit: mcg*d/mL
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2
Number analyzed (Participants) | 12 | 13 | 13 | 9 | 9
mcg*d/mL | 2672 [1700 to 3661] | 4435 [3544 to 6374] | 6654 [4040 to 8120] | 9825 [5594 to 12487] | 8639 [6159 to 12879]

6. Primary Outcome: Pharmacokinetics (PK) Parameter: Area Under the Curve (AUC) for Dose Group 5
Description: The Overall Number of Participants Analyzed represents infants. PK parameters were determined from plasma concentration-time profiles using noncompartmental methods (SAS 9.4, Cary, NC). AUC0-84 days (area-under-the-curve from 0 to 84 days) were determined using the linear trapezoidal rule. Median and range were summarized.
Time Frame: Dose Group 5 - Cohort 1: at days 0, 1, 3, 7, 14, 28; Cohort 2: at days 0, 1, 3, 7, 14, 28, 84.
Population: Participants who received the correct dose and were evaluated for PK at the designated timepoints.
Measure: Median (Full Range); unit: mcg*d/mL
Arm/Group | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 10 | 10
mcg*d/mL | 5358 [4180 to 8835] | 4462 [2840 to 6044]

7. Primary Outcome: Pharmacokinetics (PK) Parameter: Concentration for Dose Groups 1, 2, 3 and 4
Description: The Overall Number of Participants Analyzed represents infants. PK parameters were determined from plasma concentration-time profiles using noncompartmental methods (SAS 9.4, Cary, NC). Median and range were summarized for C28 days (concentration at 28 days) for Dose Groups 1, 2 and 3 and C84 days for Dose Group 4.
Time Frame: as for outcome 5
Population: Infants who received the correct dose and were evaluated for PK at the designated timepoints.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2
Number analyzed (Participants) | 12 | 13 | 13 | 9 | 9
mcg/mL | 39.19 [16.71 to 76.56] | 75.25 [47.61 to 122.59] | 124.24 [62.16 to 180.22] | 44.64 [30.83 to 64.22] | 49.60 [23.96 to 62.13]

8. Primary Outcome: Pharmacokinetics (PK) Parameter: Concentration for Dose Group 5
Description: The Overall Number of Participants Analyzed represents infants. PK parameters were determined from plasma concentration-time profiles using noncompartmental methods (SAS 9.4, Cary, NC). Median and range were summarized for C84 days (concentration at 84 days).
Time Frame: Dose Group 5 - Cohort 1: at days 0, 1, 3, 7, 14, 28; Cohort 2: at days 0, 1, 3, 7, 14, 28, 84.
Population: Participants who received the correct dose and were evaluated for PK at the designated timepoints.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 9 | 8
mcg/mL | 15.81 [11.90 to 21.42] | 19.07 [9.48 to 36.63]

9. Secondary Outcome: Percentage of Participants Who Died After Last Immunization for Dose Groups 1, 2, 3 and 4
Description: The Overall Number of Participants Analyzed represents infants. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Data for Dose Groups 1, 2, 3 and 4 are presented here.
Time Frame: From four weeks after the participants' last immunization to the end of the study follow-up (at week 48 for Dose Groups 1 and 2 and at week 96 for Dose Group 3 and 4).
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11
percentage of participants | 0 [0 to 21] | 0 [0 to 19] | 0 [0 to 21] | 0 [0 to 26] | 0 [0 to 24]

10. Secondary Outcome: Percentage of Participants Who Died After Last Immunization for Dose Group 5
Description: The Overall Number of Participants Analyzed represents infants. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated.
Time Frame: From four weeks after the participants' last immunization to the end of the study follow-up (at week 96 for Dose Group 5).
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 11 | 11
percentage of participants | 0 [0 to 24] | 0 [0 to 24]

11. Secondary Outcome: Percentage of Participants With an Occurrence of at Least One Grade 3 or Higher Adverse Event (AE) After Last Immunization for Dose Groups 1, 2, 3 and 4
Description: The Overall Number of Participants Analyzed represents infants. AE severity grading was based on the Division of AIDS (DAIDS) AE Grading table, Corrected Version 2.1. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Data for Dose Groups 1, 2, 3 and 4 are presented here.
Time Frame: From four weeks after the participants' last immunization to the end of the study follow-up (at week 48 for Dose Groups 1 and 2 and at week 96 for Dose Groups 3 and 4).
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11
percentage of participants | 23 [7 to 49] | 0 [0 to 19] | 0 [0 to 21] | 20 [4 to 51] | 18 [3 to 47]

12. Secondary Outcome: Percentage of Participants With an Occurrence of at Least One Grade 3 or Higher Adverse Event (AE) After Last Immunization For Dose Group 5
Description: The Overall Number of Participants Analyzed represents infants. AE severity grading was based on the Division of AIDS (DAIDS) AE Grading table, Corrected Version 2.1. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated.
Time Frame: as for outcome 10
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 11 | 11
percentage of participants | 18 [3 to 47] | 27 [8 to 56]

13. Secondary Outcome: Percentage of Participants With at Least One VRC01-, VRC01LS-, or VRC07-523LS-related Grade 3 or Higher Adverse Event (AE) After Last Immunization For Dose Groups 1, 2, 3, and 4
Description: The Overall Number of Participants Analyzed represents infants. AE severity grading was based on the Division of AIDS (DAIDS) AE Grading table, Corrected Version 2.1. The study sites assessed if AEs were related to study treatment. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Data for Dose Groups 1, 2, 3 and 4 are presented here.
Time Frame: as for outcome 11
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2
Number analyzed (Participants) | 13 | 14 | 13 | 10 | 11
percentage of participants | 0 [0 to 21] | 0 [0 to 19] | 0 [0 to 21] | 0 [0 to 26] | 0 [0 to 24]

14. Secondary Outcome: Percentage of Participants With at Least One VRC01-, VRC01LS-, or VRC07-523LS-related Grade 3 or Higher Adverse Event (AE) After Last Immunization for Dose Group 5
Description: The Overall Number of Participants Analyzed represents infants. AE severity grading was based on the Division of AIDS (DAIDS) AE Grading table, Corrected Version 2.1. The study sites assessed if AEs were related to study treatment. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated.
Time Frame: as for outcome 10
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 11 | 11
percentage of participants | 0 [0 to 24] | 0 [0 to 24]

15. Secondary Outcome: Percentage of Participants Diagnosed With HIV Infection After Last Immunization for Dose Groups 1, 2, 3, and 4
Description: The Overall Number of Participants Analyzed represents infants. Diagnosis testing was performed using a HIV-1 NAT (nucleic acid testing) by a method that detects DNA. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated. Data for Dose Groups 1, 2, 3 and 4 are presented here.
Time Frame: as for outcome 11
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2
Number analyzed (Participants) | 13 | 14 | 10 | 11 | 11
percentage of participants | 0 [0 to 21] | 0 [0 to 19] | 0 [0 to 21] | 0 [0 to 26] | 0 [0 to 24]

16. Secondary Outcome: Percentage of Participants Diagnosed With HIV Infection After Last Immunization for Dose Group 5
Description: The Overall Number of Participants Analyzed represents infants. Diagnosis testing was performed using a HIV-1 NAT (nucleic acid testing) by a method that detects DNA. Two-sided 90% exact Clopper-Pearson confidence intervals (CI) were calculated.
Time Frame: as for outcome 10
Population: All infants enrolled in these Dose Groups.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 11 | 11
percentage of participants | 0 [0 to 24] | 0 [0 to 24]

17. Secondary Outcome: Number of Participants Who Developed Anti-VRC Antibodies
Description: The Overall Number of Participants Analyzed represents infants with samples collected and tested. The number of infants who developed anti antibodies to the study products are summarized. For Dose Groups 1, 2, and 3, these are anti-VRC01 antibodies. For Dose Group 4, these are anti-VCR07 antibodies and for Dose Group 5, these are anti-VRC07-523LS antibodies.
Time Frame: At weeks 24 and 48.
Population: Infant study participants with samples collected and tested.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
Number analyzed (Participants) | 13 | 12 | 13 | 8 | 10 | 8 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From study entry to study completion at week 48 for Dose Groups 1 and 2 and at week 96 for Dose Groups 3, 4, and 5.
Description: Reactogenicity AEs, all grade 2 AEs assessed as possibly, probably or definitely related to the study product, and all AEs grade 3 or higher, were only collected for infants, throughout the study. Grade 1 AEs (other than reactogenicity) or grade 2 AEs not related to study product were collected until 30 days after the final immunization. AE severity grading was based on DAIDS AE Grading Table, Corrected Version 2.1. Serious adverse events (SAE) were reported according to DAIDS EAE Manual V2.0.
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 4, Cohort 1 | Dose Group 4, Cohort 2 | Dose Group 5, Cohort 1 | Dose Group 5, Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14 | 0/13 | 0/10 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/13 | 1/14 | 0/13 | 2/10 | 0/11 | 6/11 | 1/11
Other Adverse Events (participants affected / at risk) | 13/13 | 13/14 | 13/13 | 9/10 | 11/11 | 11/11 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group 1 (N=13) | Dose Group 2 (N=14) | Dose Group 3 (N=13) | Dose Group 4, Cohort 1 (N=10) | Dose Group 4, Cohort 2 (N=11) | Dose Group 5, Cohort 1 (N=11) | Dose Group 5, Cohort 2 (N=11)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
ABO haemolytic disease of newborn (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group 1 (N=13) | Dose Group 2 (N=14) | Dose Group 3 (N=13) | Dose Group 4, Cohort 1 (N=10) | Dose Group 4, Cohort 2 (N=11) | Dose Group 5, Cohort 1 (N=11) | Dose Group 5, Cohort 2 (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia neonatal (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neonatal tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Congenital pigmentation disorder (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 1 | 3 | 5 | 1 | 0 | 0 | 4
Naevus flammeus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sickle cell trait (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Strabismus congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 3 | 4 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coating in mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation neonatal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 2 | 0 | 0 | 0 | 0
Diarrhoea neonatal (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Infantile vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Regurgitation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 0 | 1 | 0
Crying (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug withdrawal syndrome neonatal (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fever neonatal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 2 | 1 | 1 | 0 | 2 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Candida nappy rash (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neonatal candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ophthalmia neonatorum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 3 | 2 | 1 | 3 | 0 | 2 | 3
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pustule (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 3 | 0 | 4 | 0 | 4 | 3
Blood albumin decreased (Investigations) | 3 | 2 | 1 | 1 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Blood bicarbonate (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 4 | 5 | 0 | 1 | 0 | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 3 | 3 | 2 | 0 | 0
Blood calcium increased (Investigations) | 3 | 4 | 0 | 2 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 3 | 2 | 1 | 2 | 1 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 5 | 6 | 0 | 2 | 0 | 3 | 0
Blood sodium decreased (Investigations) | 3 | 5 | 0 | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Capillary nail refill test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 3 | 1 | 1 | 1 | 1 | 0
Faecal volume decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 3 | 11 | 7 | 11 | 6 | 6
Liver palpable (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 4 | 3 | 6 | 4 | 7 | 2 | 3
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urine output decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Growth failure (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation neonatal (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fontanelle bulging (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infant irritability (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor neonatal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Caput succedaneum (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 2 | 2 | 0 | 0 | 0
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Poor weight gain neonatal (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decrease neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 1 | 4 | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Selective eating disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital macule (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Genital swelling (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penile rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Perineal erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal dermatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 9 | 0 | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 1 | 0
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Irregular breathing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 6 | 1 | 2 | 1 | 3
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 0 | 2 | 0 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Erythema toxicum neonatorum (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2 | 0 | 1 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Milia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 6 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash neonatal (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 1 | 4 | 0 | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient neonatal pustular melanosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT02256631/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT02256631/SAP_001.pdf